CLINICAL TRIAL: NCT01930097
Title: An Open-label, Randomized, Three-way, Cross-over Study to Compare the Efficacy of Closed-loop Operation Combined With Meal-and-carbohydrate-announcement Closed-loop Operation Combined With Meal-announcement, and Conventional Pump Therapy in Regulating Glucose Levels in Adults With Type 1 Diabetes
Brief Title: Closed-loop Control of Glucose Levels After Meal Intake in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-05
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycemia; Insulin; Glucagon; Closed-loop system; Artificial pancreas; Carbohydrate counting
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHO-dependant bolus (Active Comparator): An insulin bolus dependant of carbohydrate content will be given after each meal.
  Each subject insulin-to-carbohydrate ratio (U per 10g CHO) will be used to calculate the insulin bolus to be given. The dual-hormone closed-loop strategy will give the remaining insulin needed based on the sensor readings.
  Interventions: Other: 14 hours intervention
- CHO-independent bolus (Active Comparator): An insulin bolus independent of carbohydrate content will be given after each meal. The dual-hormone closed-loop strategy will give the remaining insulin needed based on the sensor readings.
  Interventions: Other: 14 hours intervention
- Conventional treatment (Active Comparator): Patients will use conventional pump therapy to regulate glucose levels
  Interventions: Other: 14 hours intervention

INTERVENTIONS:
Other: 14 hours intervention — Subjects will be admitted at the IRCM at 6:30. Subjects will be asked to fast from midnight. At 8:00, a standardized (50g CHO for males; 30g CHO for females) meal will be served. At 12:00, a standardized (120g CHO for males; 90g CHO for females) meal will be served. At 17:00, a standardized (70g CHO for males; 50g CHO for females) meal will be served. Between meals, patients will be allowed to do sedentary activities (reading, watching television, and playing video games, etc).

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosage based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormones: insulin and glucagon.

The objective of this project is to assess whether a dual-hormone closed-loop strategy would alleviate the burden of carbohydrate counting from patients with type 1 diabetes (T1D) without a significant degradation in post-meal glucose control.

Our primary hypothesis is that meal-announcement strategy (pre-meal CHO-independent bolus) is equivalent to meal-and-carbohydrate-announcement strategy (full CHO-matching bolus) during closed-loop regulation of glucose levels in adults with T1D. Our secondary hypothesis is that closed-loop strategy with meal-announcement strategy (pre-meal CHO-independent bolus) or meal-and-carbohydrate-announcement strategy (full CHO-matching bolus) is better than conventional pump treatment in regulation of glucose levels in adults with T1D.

DETAILED DESCRIPTION:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormone: insulin and glucagon.

Each patient will be admitted three times to a clinical research facility. In the meal-and-carbohydrate-announcement visit, patients will eat 3 meals accompanied with a matching insulin bolus (depending on the carbohydrate content of the meal) and glucose levels will be subsequently regulated using dual-hormone closed-loop system. In the meal-announcement visit, patients will eat the 3 same meals but will inject only a partial insulin bolus (not depending on carbohydrate content of the meal) and the remaining needed insulin will be delivered based on glucose sensor excursions as part of closed-loop operation. In the control visit, patients will use conventional pump therapy to regulate glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of old.
* Clinical diagnosis of type 1 diabetes for at least one year.
* The subject will have been on insulin pump therapy for at least 3 months.
* Last (less than 3 months) HbA1c ≤ 12%.

Exclusion Criteria:

* Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
* Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
* Ongoing pregnancy.
* Severe hypoglycemic episode within two weeks of screening.
* Medication likely to affect with the interpretation of the results because of their well known impact on gastric emptying: Motilium®, Prandase®, Victoza®, Byetta® and Symlin®.
* Known or suspected allergy to the trial products, meal contents including nuts, peanuts, dairy products or eggs.
* Unusual nutritional habits (e.g. vegetarians)
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
* Failure to comply with team's recommendations (e.g. not willing to eat snack, not willing to change pump parameters, etc).
* Unreliable carbohydrate counting or lack of insulin to carbohydrate ratios
* Problems with venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The positive incremental area under the curve of postprandial glucose excursions | 4 hours after meal intake
  The positive incremental area under the curve (IAUC, as compared to pre-meal glucose value) of the 4-hr postprandial glucose excursions for the breakfast, lunch and dinner meals.

SECONDARY OUTCOMES:
Mean plasma glucose | 8h00 to 21h00
Incremental two hours postprandial glucose | 2 hours after meal intake
Incremental postprandial peak-glucose values | 8h00 to 21h00
Percentage of time of plasma glucose levels between 4.0 and 10.0 mmol/L | 8h00 to 21h00
Percentage of time of plasma glucose levels spent above 10.0 mmol/L | 8h00 to 21h00
Percentage of time of plasma glucose levels spent below 4.0 mmol/L | 8h00 to 21h00
Total insulin delivery | 8h00 to 21h00
Total glucagon delivery | 8h00 to 21h00
Standard deviation of glucose levels | 8h00 to 21h00
Percentage of time of plasma glucose concentrations below 3.5 mmol/L | 8h00 to 21h00
Percentage of time of plasma glucose concentrations above 14 mmol/L | 8h00 to 21h00
Mean plasma insulin concentration | 8h00 to 21h00
Mean plasma glucagon concentration | 8h00 to 21h00
Number of patients experiencing hypoglycemia requiring oral treatment | 8h00 to 21h00
Incremental area under the curve of the 4-hr postprandial glucose excursions but the reference glucose is set to 5.0 mmol/L if premeal glucose is less than 5.0 mmol/L. | 4 hours after meal intake

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Gingras V, Rabasa-Lhoret R, Messier V, Ladouceur M, Legault L, Haidar A. Efficacy of dual-hormone artificial pancreas to alleviate the carbohydrate-counting burden of type 1 diabetes: A randomized crossover trial. Diabetes Metab. 2016 Feb;42(1):47-54. doi: 10.1016/j.diabet.2015.05.001. Epub 2015 Jun 10. PMID 26072052